CLINICAL TRIAL: NCT03614117
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Effect of a Probiotic on Recurrent Acute Otitis Media (rAOM) in Children
Brief Title: Effect of a New Probiotic Strain on Recurrent Acute Otitis Media in Children (PROMAR)
Acronym: PROMAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ProbiSearch SL (Industry)
Collaborators: Casen Recordati S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OTR/17.01
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Acute Otitis Media
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Intervention Model Description: This is an interventional, randomized, double-blind, placebo-controlled, parallel-group study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- L.salivarius PS7 6-months (Active Comparator): Lactobacillus salivarius PS7 during 6-months; approximately 1*10E9 colony forming unit (CFU) of L. salivarius PS7 in 1 sachet per day to be diluted in water by mouth for 6-months.
  Interventions: Dietary Supplement: Lactobacillus salivarius PS7 during 6 months
- L. salivarius PS7 + placebo (3+3) (Active Comparator): Lactobacillus salivarius PS7 during 3 months; approximately 1*10E9 CFU of L. salivarius PS7 in 1 sachet per day to be diluted in water by mouth for 3-months followed by 3 months oral administration of 1sachet per day of placebo supplement to be diluted in water.
  Interventions: Dietary Supplement: Lactobacillus salivarius PS7 during 3 months
- Control group (Placebo Comparator): Placebo supplement in 1 sachet per day to be diluted in water by mouth for 6-months.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus salivarius PS7 during 6 months — 7 months intervention study: A 6 months intervention period and 1 month follow-up after intervention finishing time. During the 6 months of intervention the participants will intake one daily dose of the product that contains 1*10E9 CFU of L. salivarius PS7. Then, a 1 month follow-up period will be completed.
  Other Names: Lactobacillus salivarius CECT9422 during 6 months
  Arms: L.salivarius PS7 6-months
Dietary Supplement: Lactobacillus salivarius PS7 during 3 months — 7 months intervention study: A 6 months intervention period and 1 month follow-up after intervention finishing time. During the 3 months of intervention the participants will intake one daily dose of the product that contains 1*10E9 CFU of L. salivarius PS7. After that, the participants will intake one daily dose of the placebo. Then, a 1 month follow-up period will be completed.
  Other Names: Lactobacillus salivarius CECT9422 during 3 months
  Arms: L. salivarius PS7 + placebo (3+3)
Dietary Supplement: placebo — 7 months intervention study: A 6 months intervention period and 1 month follow-up after intervention finishing time. During the 6 months of intervention the participants will intake one daily dose of placebo supplement.Then, a 1 month follow-up period will be completed.
  Arms: Control group

SUMMARY:
An interventional, randomized, double-blind, placebo-controlled study will be conducted to investigate the effect of a new probiotic strain Lactobacillus salivarius PS7 on Acute Otitis Media (AOM) in children with recurrent AOM history. The study duration will be 7 months, which includes a 6-month product administration and a 1-month follow-up period. Participants will be randomized assigned to one of the three study groups: the control group; a 3 months probiotic +3 months placebo consumption group and a 6 months probiotic consumption group. The efficacy of the probiotic strain to reduce the incidence of AOM episodes will be assessed by counting AOM episodes occurring in study participants, during the entire intervention and follow-up periods, by bilateral comparison of each of the treatment groups with the control group according to the following hypothesis: "The number of AOM episodes occurring in participants who take the probiotic is the same as that for the participants in the control group. λc = λe". Where λc is the mean incidence of AOM in the control group and λe is the mean incidence of AOM in the groups taking the probiotic strain Lactobacillus salivarius PS7 obtained with 95% confidence interval.

DETAILED DESCRIPTION:
The parent or legal guardian of the minors will be contacted during a visit to the pediatrician for suspected AOM to request their participation in the study, which will be voluntary.

The study visits will take place at the primary care center or hospital. During Visit 1, the inclusion and exclusion criteria will be verified, and the informed consent will be signed. Information will be collected on the demographic profile, characteristics of the AOM episode and the prescribed treatment; and the participants will be randomized. The investigator will give the parent or guardian the product corresponding to the first treatment period (3 months) and will explain how to administer it to the child, as well as when the next visits will take place and what they will entail. Instructions will be given to start the administration of the product as soon as possible after the collection of the first stool sample. A sample will be collected from the outer ear most affected by the AOM using a sterile swab (Day 0). The investigator will go over, with the parent or legal guardian, the details of the diary to be completed (Annex II), how to record the data on product administration, fever episodes, days of school or daycare missed, unscheduled visits to the pediatrician, as well as data related to the frequency and characteristics of the stools in the event of AOM episodes and/or antibiotic treatment. The investigator will inform the parent or legal guardian that, during the child's participation in the study, the child cannot take any probiotic supplement.

During Visit 2, a sample will be taken from the same ear as in the previous visit using a sterile swab. Any questions regarding completing the diary will be discussed. The leftover product from the first treatment period will be collected and the study product corresponding to the second supplement administration period will be dispensed.

At the third visit (Visit 3, after 6 months of product administration), a sample will be collected from the same ear as in previous visits using a sterile swab. Any leftover product from the second treatment period will be collected.

During the fourth visit (Visit 4, after 1 month of observation), a sample will be collected from the same ear as in previous visits using a sterile swab. The completed diary will be collected.

Throughout the duration of the child's participation in the study (7 months), additional visits to the pediatrician (study investigator) may take place. If an episode of AOM, otitis externa or respiratory tract infection occurs during the intervention period, the investigator will make a diagnosis and will start the necessary treatment. In the course of new AOM episodes, during the intervention period, the administration of the product will not be interrupted. If the AOM episode occurs during the observation period, the investigator will proceed according to his/her routine practice. At the additional visits taking place, relevant data will be collected on the possible Adverse Events (AEs) or Serious Adverse Events (SAEs), as well as on the concomitant medication.

ELIGIBILITY:
Inclusion Criteria:

* Children 1 to 4 years of age with rAOM (3 episodes of AOM in the last 6 months, or 4 in the last 12 months).
* Written informed consent signed by one of parents or legal guardian with the express or tacit consent of the other.
* Presence of an AOM episode at the time of inclusion in the study.

Exclusion Criteria:

* chronic conditions under regular medication, such as asthma, allergic rhinitis…
* congenital or acquired immunodeficiency,
* taking systemic corticoid in the last 3 months for longer than 1 month
* under present prophylactic antibiotic treatment
* Down syndrome,
* cleft lip or palate,
* chronic tympanic perforation,
* craniofacial abnormalities,
* sleep apnea syndrome,
* planned tympanostomy or tonsillectomy during the months of the study,
* short bowel syndrome or any surgery in the gastrointestinal tract,
* intestinal epithelial barrier defect (e.g., chronic diarrhea, intestinal inflammation),
* metabolic disorders (diabetes, etc.),
* heart failure and cardiac medical history (e.g. artificial heart valve, medical history of infective endocarditis, rheumatic fever or cardiac malformation),
* uncertainty of the investigator regarding the willingness or capacity of the parents or legal guardian of the child to comply with the requirements of the protocol.

Ages: 1 Year to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 222 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2020-07-06 (Actual); Study Completion 2020-07-06 (Actual)

PRIMARY OUTCOMES:
Number of AOM episodes | 7 months
  Number of AOM episodes suffered by participants

SECONDARY OUTCOMES:
Patients (%) with at least one AOM episode during the intervention and follow-up periods. | 7 months
  % of patients with at least one AOM episode
Number of AOM episodes after 3 months of product intake. | 3 months
  Number of AOM episodes suffered by participants after 3 months of product intake
Time from onset of first AOM episode to the onset of the next episode. | 7 months
  Number of days from onset of first AOM episode to the onset of the next episode.
Adverse events and/or serious adverse events | 7 months
  The number, duration and possible relationship of (serious) adverse events to the study product.

OTHER OUTCOMES:
Variables assessing compliance with the protocol | 7 months
  The variables assessing compliance with the protocol
  * Study product administration.
  * Probiotic supplement administration
  * Compliance with the visit/assessment intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Susana Manzano, PhD, Study Chair — ProbiSearch SL
Locations (1):
- Hospital Universitario QuirónSalud Pozuelo, Pozuelo de Alarcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided